CLINICAL TRIAL: NCT04864704
Title: Immediate Decrease of Muscle Biomechanical Stiffness Following Dry Needling in Asymptomatic Participants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bradley University (Other)
Responsible Party: Principal Investigator, Joseph Kelly, Assistant Professor, Bradley University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BradleyU
Record Dates: First submitted 2021-04-20; First posted 2021-04-29 (Actual); Last update posted 2021-04-29 (Actual); Status verified 2021-04

CONDITIONS: Healthy
MeSH Terms: interventions — Dry Needling

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Infraspinatus (Active Comparator): Subjects infraspinatus stiffness was measured and observed
  Interventions: Other: dry needling
- Erector spinae (Active Comparator): Subjects erector spinae stiffness was measured and observed
  Interventions: Other: dry needling
- Gastrocnemius (Active Comparator): Subjects gastrocnemius stiffness was measured and observed
  Interventions: Other: dry needling

INTERVENTIONS:
Other: dry needling — Physical therapy

SUMMARY:
60 healthy participants were randomized into infraspinatus, erector spinae, or gastrocnemius groups. One session of dry needling DN was applied to the muscle in standardized location. Stiffness was assessed using a MyotonPRO at baseline, immediately post DN, and 24 hours later. The presence of a localized twitch response (LTR) during DN was used to subgroup participants.

ELIGIBILITY:
Inclusion Criteria:

* men and women ages 18 to 65 years
* reported good general health
* tenderness or palpable trigger point in the muscle (infraspinatus, gastrocnemius, or erector spinae)

Exclusion Criteria:

* BMI > 30kg/m2
* surgery in the prior 12 months
* current pain in the shoulder, low back, and lower leg
* precautions to dry needling treatment (anticoagulant medications, bleeding disorders, known pregnancy)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2014-01-30 (Actual); Primary Completion 2015-01-30 (Actual); Study Completion 2015-01-30 (Actual)

PRIMARY OUTCOMES:
Change in Stiffness | Change from baseline and immediately post intervention
  Biomechanical stiffness of the muscle measured, non-invasively using a MyotonPRO. Stiffness (N/m)

CONTACTS AND LOCATIONS:
Locations (1):
- Bradley University, Peoria, Illinois, United States

IPD SHARING:
Plan to Share IPD: No
Data will not be shared